CLINICAL TRIAL: NCT00004445
Title: Eight Channel Implanted Neuroprosthesis for Exercise, Standing and Transfers
Brief Title: Study of an Implantable Functional Neuromuscular Stimulation System for Patients With Spinal Cord Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Ronald J. Triolo, Biomedical Enginer, Case Western Reserve University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 199/13455; CWRU-FDR001244 (Other Grant/Funding Number: US FDA Offoce of Orphan product Development)
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Results first posted 2019-07-22 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Spinal Cord Injury
Keywords: environmental/toxic disorders; neurologic and psychiatric disorders; rare disease; spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Implanted Neuroprosthesis (Experimental): Volunteers are evaluated for appropriateness for inclusion in the study on an intent-to-treat basis. Qualifying candidates all receive the implanted neuroprosthesis and participate in post-operative training and follow-up procedures.
  Interventions include:
  Procedure/Surgery Rehabilitation/Exercise
  Device includes:
  IRS-8 Stimulating Electrodes External Controller
  Interventions: Procedure: Surgery; Device: IRS-8

INTERVENTIONS:
Procedure: Surgery
Device: IRS-8

SUMMARY:
OBJECTIVES:

I. Establish the procedures for implementing and assessing the clinical utility of functional neuromuscular stimulation using an implanted eight-channel standing and transfer system in patients with incomplete tetraplegia or paraplegia.

II. Develop and apply quantitative functional evaluations of system performance in these patients.

III. Perform long term follow up and monitor system use outside of the laboratory.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients undergo surgery in which electrodes are sutured into areas of the pelvis and legs. Electrode leads are inserted into a receiver/stimulator implanted in a subcutaneous pocket in the abdomen. Following implantation, patients undergo training in standing, transfers, and other advanced mobility skills using the functional neuromuscular stimulation system. Restricted activity continues for 2 weeks after surgery, followed by 8 weeks of exercise. Standing training then begins, and continues for up to 6 weeks. Home-based training follows prior to discharge with the system for spontaneous use.

Patients are followed at 3, 6, and 12 months, then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

Low cervical or thoracic spinal cord injuries (C6-T12) Must be skeletally mature ASIA impairment scale A (complete motor and sensory deficits), B (sensory sparing), or C (motor and sensory sparing) Intact lower motor neurons Greater than 6 months since injury Range of motion within normal limits No renal compromise No cardiac abnormalities No circulatory compromise No pulmonary compromise No acute or chronic psychological problems or chemical dependency No acute orthopedic complications (scoliosis, history of spontaneous fractures, dislocations, etc.) No acute medical complications (no skin breakdowns, uncontrolled seizures, immunological compromise, etc.)

Exclusion Criteria:

Failure to meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 1996-09; Primary Completion 2009-09 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald J. Triolo, Study Chair — Case Western Reserve University
Locations (2):
- United States (2):
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth System, Cleveland, Ohio

REFERENCES:
- [Derived] Triolo RJ, Bailey SN, Foglyano KM, Kobetic R, Lombardo LM, Miller ME, Pinault G. Long-Term Performance and User Satisfaction With Implanted Neuroprostheses for Upright Mobility After Paraplegia: 2- to 14-Year Follow-Up. Arch Phys Med Rehabil. 2018 Feb;99(2):289-298. doi: 10.1016/j.apmr.2017.08.470. Epub 2017 Sep 9. PMID 28899825
- [Derived] Rohde LM, Bonder BR, Triolo RJ. Exploratory study of perceived quality of life with implanted standing neuroprostheses. J Rehabil Res Dev. 2012;49(2):265-78. doi: 10.1682/jrrd.2010.08.0156. PMID 22773528
- [Derived] Triolo RJ, Bailey SN, Miller ME, Rohde LM, Anderson JS, Davis JA Jr, Abbas JJ, DiPonio LA, Forrest GP, Gater DR Jr, Yang LJ. Longitudinal performance of a surgically implanted neuroprosthesis for lower-extremity exercise, standing, and transfers after spinal cord injury. Arch Phys Med Rehabil. 2012 May;93(5):896-904. doi: 10.1016/j.apmr.2012.01.001. PMID 22541312

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of participants is based on evaluation of past medical history and in person evaluation including strength, ROM, and response to stimulation to determine eligibility.
Pre-assignment Details: Participants will go through a screening process that will determine eligibility for the study. If they don't meet the inclusion or exclusion criteria they will not be invited to continue to the second phase of the study.
Groups:
- Implanted Neuroprosthesis: Volunteers are evaluated for appropriateness for inclusion in the study on an intent-to-treat basis. Qualifying candidates all receive the implanted neuroprosthesis and participate in [ost-operative training and follow-up procedures.
  Surgery
  IRS-8
Period: Overall Study
Arm/Group | Implanted Neuroprosthesis
Started | 18
Completed | 15
Not Completed | 3
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Implanted Neuroprosthesis
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Standing Performance
Description: A measure of how long an individual can maintain a standing position.
Time Frame: Discharge, 1 follow-up between 6-12 months follow-up
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Implanted Neuroprosthesis: Volunteers are evaluated for appropriateness for inclusion in the study on an intent-to-treat basis. Qualifying candidates all receive the implanted neuroprosthesis and participate in post-operative training and follow-up procedures.
  Interventions include:
  Procedure/Surgery Rehabilitation/Exercise
  Device includes:
  IRS-8 Stimulating Electrodes External Controller
  Surgery
  IRS-8
Arm/Group | Implanted Neuroprosthesis
Number analyzed (Participants) | 15
minutes
  Discharge standing time | 27.4 (38.6)
  6-12 month follow-up standing time | 15.6 (21.8)

2. Secondary Outcome: Distribution of Body Weight Through the Legs and Arms While Standing
Description: Measure of how much weight is placed on the legs and arms while standing
Time Frame: Discharge, 1 follow-up between 6-12 months
Measure: Mean (Standard Deviation); unit: percentage of body weight
Arm/Group | Implanted Neuroprosthesis
Number analyzed (Participants) | 15
percentage of body weight
  Discharge body weight distribution | 90.0 (13.1)
  6-12 month follow-up body weight distribution | 76.7 (22.2)

ADVERSE EVENTS:
Arm/Group | Implanted Neuroprosthesis
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implanted Neuroprosthesis (N=15)
Infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No